CLINICAL TRIAL: NCT04033640
Title: Evaluation of a Diagnostic to Identify G6PD Deficiency in Brazil
Brief Title: Evaluation of a Diagnostic to Identify Glucose-6-phosphate Dehydrogenase (G6PD) Deficiency in Brazil
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: PATH (Other)
Collaborators: Fundação de Medicina Tropical Dr. Heitor Vieira Dourado (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: G6PD Brazil
Record Dates: First submitted 2019-07-17; First posted 2019-07-26 (Actual); Results first posted 2021-11-11 (Actual); Last update posted 2021-11-11 (Actual); Status verified 2021-09

CONDITIONS: G6PD Deficiency
Keywords: G6PD deficiency
MeSH Terms: conditions — Glucosephosphate Dehydrogenase Deficiency | interventions — Blood Cell Count

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- G6PD Diagnostic Testing (Other): Participants provided whole blood samples as well as finger-stick capillary blood samples.
  At the clinic site, study staff performed the SD Biosensor STANDARD G6PD test and the POC HemoCue hemoglobin test on finger stick blood samples.
  At the reference laboratories, G6PD activity was measured from whole blood samples using the SD Biosensor STANDARD G6PD test and the Pointe Scientific G6PD reference assay and hemoglobin was measured using the HemoCue hemoglobin test and by a complete blood count (CBC) using an automated hematology analyzer (Manaus site only).
  Interventions: Diagnostic Test: SD Biosensor STANDARD G6PD Test; Diagnostic Test: Pointe Scientific Test Kit; Diagnostic Test: HemoCue System; Diagnostic Test: Complete blood count (CBC)
- Health Workers (No Intervention): Participants were trained on use of the SD Biosensor STANDARD G6PD test by members of the study team with extensive experience with G6PD diagnostics and the STANDARD G6PD test. Health worker participants were surveyed to assess label and packing comprehension as well as results interpretation.

INTERVENTIONS:
Diagnostic Test: SD Biosensor STANDARD G6PD Test — The SD Biosensor G6PD Analyzer is designed to measure the quantitative determination of total hemoglobin concentration and G6PD enzymatic activity in fresh human whole blood specimens based on reflectometry assays in a point-of-care (POC) setting. The test is intended to aid in the identification of people with G6PD deficiency.
  The test is currently not licensed for use in Brazil and is considered an investigational product.
  Arms: G6PD Diagnostic Testing
Diagnostic Test: Pointe Scientific Test Kit — The Pointe Scientific test kit will serve as the reference assay to assess G6PD activity. Its intended use is for the quantitative, kinetic determination of G6PD in blood at 340 nm.
  Arms: G6PD Diagnostic Testing
Diagnostic Test: HemoCue System — The HemoCue hemoglobin (Hb) 201+ system is designed for quantitative point-of-care whole blood hemoglobin determination in primary care using a specially designed analyzer, the HemoCue Hb 201+ Analyzer, and specially designed microcuvettes, the HemoCue Hb 201+Microcuvettes.
  Arms: G6PD Diagnostic Testing
Diagnostic Test: Complete blood count (CBC) — In Manaus, hemoglobin concentration was determined by CBC using an automated hematology analyzer (Sysmex KX-21N).
  Arms: G6PD Diagnostic Testing

SUMMARY:
Th objectives of this study are:

* To determine the performance of G6PD tests in detecting G6PD activity and hemoglobin (Hb) compared to a reference assay
* To assess the comprehension of the G6PD test packaging and labelling among intended users
* To assess the usability of G6PD test result outputs among intended users

DETAILED DESCRIPTION:
This is a cross-sectional diagnostic accuracy study that includes both participants and health worker participants.

The participant population will be recruited at clinics and through a household survey using an enriched sample of a population with known G6PD status, established through previous epidemiological studies. Clinic staff will take capillary blood samples and conduct two point of care (POC) tests: 1) HemoCue® hemoglobin test, and 2) the investigational Standard Diagnostics (SD) Biosensor STANDARD POC test for glucose-6-phosphate dehydrogenase (G6PD) deficiency. Venous blood will be collected and transferred to a laboratory where reference assays will be performed on venous samples using the Pointe Scientific G6PD Analyzer and hemoglobin tests.

The health worker participants will include trained intended users of the G6PD tests. Trained health workers will be surveyed to assess product usability through a questionnaire to assess label and packing comprehension as well as results interpretation.

ELIGIBILITY:
1. Participants with unknown G6PD status

   Inclusion criteria:
   * Febrile patients seeking care at the Manaus or Porto Velho clinics
   * 2 years age or older
   * Willing to provide informed consent

   Exclusion criteria
   * Younger than 2 years of age
   * Participants who received a blood transfusion in the last 3 months, self report
   * Unwilling to provide informed consent
2. Participants with known G6PD status

   Inclusion criteria:
   * Included in previous G6PD surveys and provided consent to be contacted again
   * 2 years of age or older
   * Willing to provide informed consent or assent

   Exclusion criteria:
   * Younger than 2 years of age
   * Participants who received a blood transfusion in the last 3 months, self report
   * Unwilling to provide informed consent or assent or unavailable during study visit
3. Health workers

Inclusion Criteria:

* Provides malaria case management at study facility or study site
* Considered an intended user of quantitative POC G6PD tests
* Trained and proficient in the use of the POC G6PD test
* Willing to provide informed consent

Exclusion Criteria:

* Does not provide malaria case management at study facility or study site
* Not considered an intended user of quantitative POC G6PD tests
* Not trained or not proficient in the use of the POC G6PD test
* Unwilling to provide informed consent

Min Age: 2 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 1754 (Actual)
Dates: Start 2019-06-27 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2019-12-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Marcus Lacerda, MD, PhD, Principal Investigator — FMT/HVD
Locations (2):
- Brazil (2):
  - Tropical Medicine Foundation Doctor Heitor Vieira Dourado, Manaus, Amazonas
  - Centro de Pesquisa em Medicina Tropical de Rondônia, Porto Velho, Rondônia

IPD SHARING:
Plan to Share IPD: No
There is no plan to share any IPD with other researchers.

REFERENCES:
- [Derived] Zobrist S, Brito M, Garbin E, Monteiro WM, Clementino Freitas S, Macedo M, Soares Moura A, Advani N, Kahn M, Pal S, Gerth-Guyette E, Bansil P, Domingo GJ, Pereira D, Lacerda MV. Evaluation of a point-of-care diagnostic to identify glucose-6-phosphate dehydrogenase deficiency in Brazil. PLoS Negl Trop Dis. 2021 Aug 12;15(8):e0009649. doi: 10.1371/journal.pntd.0009649. eCollection 2021 Aug. PMID 34383774
- [Derived] Gerth-Guyette E, Adissu W, Brito M, Garbin E, Macedo M, Sharma A, Das S, Lacerda MVG, Pereira D, Talukdar A, Yilma D, Pal S, Zobrist S, Domingo GJ. Usability of a point-of-care diagnostic to identify glucose-6-phosphate dehydrogenase deficiency: a multi-country assessment of test label comprehension and results interpretation. Malar J. 2021 Jul 8;20(1):307. doi: 10.1186/s12936-021-03803-1. PMID 34238299

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This diagnostic accuracy study was conducted at 2 centers situated in the Brazilian Amazon and included both participants and health workers. Participants were recruited at clinics and through an enriched sample in Manaus and Porto Velho, Brazil. Health worker participants included both health care providers, such as community health workers/field agents, and laboratory technicians who perform malaria rapid diagnostic tests and other malaria testing near the point of care (POC).
Groups:
- G6PD Diagnostic Testing: Participants provided whole blood samples as well as finger-stick capillary blood samples.
  At the clinic site, study staff performed the Standard Diagnostics (SD) Biosensor STANDARD glucose-6-phosphate dehydrogenase (G6PD) test and the POC HemoCue hemoglobin test on finger stick blood samples.
  At the reference laboratories, G6PD activity was measured from whole blood samples using the SD Biosensor STANDARD G6PD test and the Pointe Scientific G6PD reference assay and hemoglobin was measured using the HemoCue hemoglobin test and by a complete blood count (CBC) using an automated hematology analyzer (Manaus site only).
- Health Workers: Participants were trained on use of the STANDARD G6PD test by members of the study team with extensive experience with G6PD diagnostics and the STANDARD G6PD test. Health worker participants were surveyed to assess label and packing comprehension as well as results interpretation.
Period: Overall Study
Arm/Group | G6PD Diagnostic Testing | Health Workers
Started | 1736 | 18
Completed | 1736 | 18
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Demographic information were not collected for the health worker participants in this study.
Groups:
- G6PD Diagnostic Testing: Participants provided whole blood samples as well as finger-stick capillary blood samples.
  At the clinic site, study staff performed SD Biosensor STANDARD G6PD test and the POC HemoCue hemoglobin test on finger stick blood samples.
  At the reference laboratories, G6PD activity was measured from whole blood samples using the SD Biosensor STANDARD G6PD test and the Pointe Scientific G6PD reference assay and hemoglobin was measured using the HemoCue hemoglobin test and by CBC.
- Total: Total of all reporting groups
Arm/Group | G6PD Diagnostic Testing | Health Workers | Total
Number analyzed (Participants) | 1736 | 18 | 1754
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: Demographic information were not collected for the health worker participants in this study.
  years
    number analyzed (Participants) | 1736 | 0 | 1736
    (all) | 37.7 (13.9) |  | 37.7 (13.9)
Age, Customized [Count of Participants; unit: Participants] — Population: Demographic information were not collected for the health worker participants in this study.
  Participants
    number analyzed (Participants) | 1736 | 0 | 1736
    2-11 years | 24 |  | 24
    12-15 years | 22 |  | 22
    16-64 years | 1632 |  | 1632
    65+ years | 58 |  | 58
Sex: Female, Male [Count of Participants; unit: Participants] — Population: Demographic information were not collected for the health worker participants in this study.
  Participants
    number analyzed (Participants) | 1736 | 0 | 1736
    Female | 948 |  | 948
    Male | 788 |  | 788
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Brazil | 1736 | 18 | 1754

OUTCOME MEASURES:

1. Primary Outcome: Sensitivity of SD Biosensor STANDARD G6PD Test for Identifying G6PD Deficient Individuals
Description: For the purposes of this study, an individual was considered G6PD deficient if they tested positive in the Pointe Scientific assay. A true positive was defined as a participant with ≤ 30% of normal G6PD activity in circulating venous blood determined by the Pointe Scientific test.
  Diagnostic sensitivity of the SD Biosensor STANDARD G6PD test is defined as the percentage of participants who tested positive for G6PD deficiency on the reference test who were identified by the test assay as positive, calculated as:
  Number of participants who were both test and true positive / (Number of participants who were test and true positive + Number of participants who were test negative but true positive [ie false negative]) * 100%.
  Sensitivity of the SD Biosensor STANDARD G6PD test was calculated from both venous and capillary blood samples.
Time Frame: All samples were collected on study day 1
Population: Participants with available data
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | G6PD Diagnostic Testing
Number analyzed (Participants) | 1693
percentage of participants
  Venous blood: number analyzed (Participants) | 1662
  Venous blood | 100.0 [93.6 to 100.0]
  Capillary blood | 100.0 [93.8 to 100.0]

2. Primary Outcome: Sensitivity of SD Biosensor STANDARD G6PD Test for Identifying Women With Intermediate G6PD Activity
Description: To investigate the performance of the SD Biosensor STANDARD G6PD test to distinguish females with intermediate G6PD activity from females with normal activity, assay sensitivity was determined at a G6PD activity threshold of 70%. A true positive for intermediate G6PD activity in females was defined as G6PD activity between 30 and 70% of normal in circulating venous blood as determined by the Pointe Scientific test.
  Sensitivity of the SD Biosensor STANDARD G6PD test is the percentage of women who tested positive for intermediate G6PD activity on the reference test who were identified by the test assay as positive, calculated as:
  Number of women who were both test and true positive / (Number of women who were test and true positive + Number of women who were test negative but true positive [ie false negative]) * 100%.
  Sensitivity of the SD Biosensor STANDARD G6PD test for identifying females with intermediate G6PD activity was calculated from both venous and capillary blood samples.
Time Frame: All samples were collected on study day 1
Population: Female participants with available data
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | G6PD Diagnostic Testing
Number analyzed (Participants) | 918
percentage of participants
  Venous blood: number analyzed (Participants) | 911
  Venous blood | 96.9 [83.8 to 99.9]
  Capillary blood | 94.3 [80.8 to 99.3]

3. Primary Outcome: Specificity of SD Biosensor STANDARD G6PD Test for Identifying G6PD Deficient Individuals
Description: For the purposes of this study, an individual was considered G6PD deficient if they tested positive by the Pointe Scientific assay. A true negative was defined as > 30% of normal G6PD activity in circulating venous blood as determined by the Pointe Scientific test.
  Specificity is the percentage of participants who tested negative for G6PD deficiency on the reference test who were identified as negative using the test assay, calculated as:
  Number of participants who were both test and true negative / (Number of participants who were test and true negative + Number of participants who were test positive but true negative [ie false positive]) * 100%.
  Specificity of the SD Biosensor STANDARD G6PD test was calculated from both venous and capillary blood samples.
Time Frame: All samples were collected on study day 1
Population: Participants with available data
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | G6PD Diagnostic Testing
Number analyzed (Participants) | 1693
percentage of participants
  Venous blood: number analyzed (Participants) | 1662
  Venous blood | 98.6 [97.9 to 99.1]
  Capillary blood | 97.8 [97.0 to 98.5]

4. Primary Outcome: Specificity of SD Biosensor STANDARD G6PD Test for Identifying Women With Intermediate G6PD Activity
Description: To investigate the performance of the SD Biosensor STANDARD G6PD test to distinguish females with intermediate G6PD activity from females with normal activity, the specificity was determined at a G6PD activity threshold of 70%. A true negative for intermediate G6PD activity in females was defined as G6PD activity > 70% of normal in circulating venous blood as determined by the Pointe Scientific test.
  Specificity is the percentage of participants who tested negative for G6PD deficiency on the reference test who were identified as negative using the test assay, calculated as: Number of participants who were both test and true negative / (Number of participants who were test and true negative + Number of participants who were test positive but true negative [ie false positive]) * 100%.
  Specificity of the SD Biosensor STANDARD G6PD test was calculated from both venous and capillary blood samples.
Time Frame: All samples were collected on study day 1
Population: Female participants with available data
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | G6PD Diagnostic Testing
Number analyzed (Participants) | 918
percentage of participants
  Venous blood: number analyzed (Participants) | 911
  Venous blood | 96.5 [95.0 to 97.6]
  Capillary blood | 92.3 [90.3 to 94.0]

5. Secondary Outcome: Accuracy Between the SD Biosensor STANDARD G6PD Test Assay and the Pointe Scientific Test Kit
Description: Accuracy between the SD Biosensor STANDARD G6PD test assay and the Pointe Scientific G6PD reference assay was calculated as the percent agreement between both G6PD tests, ie, the percentage of participants with the same diagnosis according to both tests (either deficient, intermediate, or normal G6PD levels).
  Accuracy of the SD Biosensor STANDARD G6PD test was calculated from both venous and capillary blood samples.
Time Frame: All samples were collected on study day 1
Population: Participants with available data
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | G6PD Diagnostic Testing
Number analyzed (Participants) | 1693
percentage of participants
  Venous blood: number analyzed (Participants) | 1662
  Venous blood | 96.7 [95.7 to 97.5]
  Capillary blood | 94.1 [92.9 to 95.2]

6. Secondary Outcome: Accuracy Between the SD Biosensor STANDARD G6PD Test Measure of Hemoglobin and the Reference HemoCue Hemoglobin Test
Description: Accuracy between the SD Biosensor STANDARD G6PD test measure of hemoglobin and the HemoCue hemoglobin reference assay was calculated as the percentage agreement between both tests, ie, the percentage of participants with the same diagnosis according to both tests (either non/mild anemia, moderate anemia or severe anemia).
Time Frame: All samples were collected on study day 1
Population: Participants with available data
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | G6PD Diagnostic Testing
Number analyzed (Participants) | 1693
percentage of participants
  Venous blood: number analyzed (Participants) | 1662
  Venous blood | 93.3 [92.0 to 94.5]
  Capillary blood | 91.8 [90.4 to 93.1]

7. Secondary Outcome: Accuracy Between the SD Biosensor STANDARD G6PD Test Measure of Hemoglobin and the Hemoglobin Measured in a Complete Blood Count
Description: Accuracy between the SD Biosensor STANDARD G6PD test measure of hemoglobin and the hemoglobin result from the complete blood count (CBC) reference assay (using an automated hematology analyzer) was calculated as the percentage agreement between both tests, ie, the percentage of participants with the same diagnosis according to both tests (either non/mild anemia, moderate anemia or severe anemia). Complete blood counts were only conducted for participants enrolled at the site in Manaus.
Time Frame: All samples were collected on study day 1
Population: Participants enrolled at the site in Manaus with available data
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | G6PD Diagnostic Testing
Number analyzed (Participants) | 900
percentage of participants
  Venous blood: number analyzed (Participants) | 850
  Venous blood | 93.1 [91.1 to 94.7]
  Capillary blood | 93.2 [91.4 to 94.8]

8. Secondary Outcome: Median G6PD Values Measured by the SD Biosensor STANDARD G6PD Test for Venous and Capillary Blood Samples
Time Frame: All samples were collected on study day 1
Population: Participants with available data
Measure: Median (95% Confidence Interval); unit: units / gram of hemoglobin
Arm/Group | G6PD Diagnostic Testing
Number analyzed (Participants) | 1735
units / gram of hemoglobin
  Venous blood: number analyzed (Participants) | 1713
  Venous blood | 8.0 [7.1 to 9.1]
  Capillary blood | 7.6 [6.6 to 8.8]
Statistical Analysis 1: Comparison: G6PD Diagnostic Testing; Comparison of SD Biosensor POC G6PD test results for capillary and venous samples; Test type: Other; p < 0.001, K-sample test; The p-value was calculated using a nonparametric k-sample test on the equality of medians

9. Secondary Outcome: Number of Participants Who Met Acceptance Criteria for Label Comprehension
Description: After completing training, health worker participants were asked to complete a questionnaire to assess their comprehension of the test label. The questionnaire consisted of 13 multiple-choice questions with mutually exclusive options and a single correct answer focused on aspects of the product label including key warnings, limitations, and restrictions as well as the proper test procedure.
  Acceptance (success) criterion for label comprehension was defined as at least 85% correct responses (11 out of 13 possible points).
Time Frame: Day 1
Population: Health worker participants
Measure: Count of Participants; unit: Participants
Arm/Group | Health Workers
Number analyzed (Participants) | 18
Participants | 10

10. Secondary Outcome: Number of Participants Who Met Acceptance Criteria for Accurate Results Interpretation
Description: After completing training, health worker participants were asked to complete a questionnaire to assess their ability to interpret the test result outputs. The questionnaire consisted of seven short-answer questions (5 valid results, 2 invalid results) focused on the participant's ability to read the results screen, record the simulated G6PD and hemoglobin quantitative results, and classify the results as normal, intermediate, deficient, or invalid.
  For each valid result, three points were possible: (one for G6PD result transcription, one for hemoglobin result transcription, and one for result interpretation) and for each invalid result, one point was possible, resulting in a total of 17 possible points.
  Acceptance (success) criterion for results interpretation was defined as at least 85% correct responses (15 out of 17 possible points).
Time Frame: Day 1
Population: Health worker participants
Measure: Count of Participants; unit: Participants
Arm/Group | Health Workers
Number analyzed (Participants) | 18
Participants | 16

ADVERSE EVENTS:
Time Frame: Approximately 30 minutes
Description: Health worker participants were not monitored for safety and no adverse event or mortality information were collected.
Arm/Group | G6PD Diagnostic Testing | Health Workers
All-Cause Mortality (participants affected / at risk) | 0/1736 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/1736 | 0/0
Other Adverse Events (participants affected / at risk) | 0/1736 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-05-05): https://cdn.clinicaltrials.gov/large-docs/40/NCT04033640/Prot_SAP_000.pdf